CLINICAL TRIAL: NCT04613336
Title: Efficacy of Topical Heparin Spray on Donor Site Wound Healing Time Compared to Conventional Dressing Among Patients Undergoing Split Thickness Skin Grafting
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Faraz Adil, Principal Investigator, Dow University of Health Sciences
Other Study IDs: dow123
Record Dates: First submitted 2020-10-16; First posted 2020-11-03 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Wound Healing

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Wound is defined by the breach in dermis of the skin. It can be caused by road traffic accidents, tumor excision, chronic illness like diabetes, bed sores in bedridden patients, burns, insects' bites etc. Treatment goals for wound coverage includes earliest debridement, dressings, local antibiotics, limb elevation, fracture fixations and wound coverage. Skin graft functions both as occlusive dressing, as a skin replacement and as a stimulus for healing. Even though the usage of flaps to cover the wounds has been increased recently still skin grafting serves as an easiest and simplest way of covering the wound. However, skin grafting introduces another wound in addition to the existing wound, the donor site wound (DSW). A secondary donor-site wound (DSW) is formed after harvesting split thickness skin graft which adds up with the primary wound to increase the total size of the wounds for the healing process. This donor site wound cause itching, pain and cosmetic embarrassment. That is why the proper and timely healing of the donor site wound is of great importance. Basic management of DSWs includes conventional dressings that provides absorption of bleeding solely.

DETAILED DESCRIPTION:
This is a randomized control trial that will be conducted at Dr. Ruth K.M. Pfau, Civil Hospital Karachi for a duration of six months after approval of the synopsis. Randomization will be done using sequentially numbered, opaque, sealed envelopes (SNOSE). A sample size of total 60 patients was calculated through OpenEpi. Patients will be counseled about the procedure of grafting and change of dressings postoperatively. Inclusion Criteria: age between 18 to 55 years, both genders, non-hypertensive patients, hemoglobin levels more than 10 g/dl, Platelet count above 150 to 400 × 109/L, wounds for more than 6 weeks. Exclusion Criteria: Hypertensive patients, bleeding tendencies (Disorder), immune-compromised, familial history of bleeding. The trial will be registered with clinical trial unit (CTU) of the Dow University of Health Sciences. Statistical analyses will be done using SPSS version 21. Descriptive analyses will be reported for all variables including age, gender, treatment group distribution and other independent and dependent variables. Inferential statistics will be reported using comparison of treatment groups using repeated measure ANOVA. P-value of <0.05 will be considered as significant. The expected total expenditure on the research project will be twenty thousand.

Data will be collected with change of dressings at graft donor site wound (DSW) that is the thigh. Study objectives will be discussed and explained to the patients before surgery as part of their change of dressings post operatively as in routine. Potential benefits and discomforts of the procedure will be explained. There is no potential adverse effects of heparin on wound or patients. Participants will receive both oral and written information about the study. Consent form will be filled by the participants. Questionnaire with photographic assessment will be filled at every change of dressing.

Split-thickness skin graft will be harvested from medial side of thigh in two strips of about 10*6cm with a few cm break in between them, with a Humby knife adjusted on with a randomized setting to harvest a fixed depth of skin graft. After harvesting the graft the donor site wound will be photographed, cleaned with saline and dressed with impregnated wax gauzes and sterilized cotton covered in roll gauze.

At first postoperative day, donor site cotton dressing will be opened. Heparin and conventional dressing group allocation will be done through randomization in order to prevent any confounding factors such as baseline differences in depth of wound. Patients will be provided with paper chits to choose from, with A or B marked on it. The proximal strip of donor site wound (DSW) will be dressed according to the chit chosen. Patients picking up A chit will be dealt as 'control half (conventional dressing)', where by patients picking up B chit will be dealt as 'intervention half'.

The 'control half' will be redressed with sterilized cotton covered in roll gauze whereas 'intervention half' of wound will be sprayed with 5000 I.U/ml concentration of the heparin placed in a 5 cc syringe. Then the wound will be redressed with sterilized cotton covered in roll gauze. This will be repeated on donor site 'intervention half' of wound on daily basis.

Skin graft donor site wound will be inspected by the faculty of Plastic surgery on the 7th post-operative day and photographic assessment will be recorded.

The visual analogue scale (VAS) will be used to access pain

Wound healing will be assessed by following parameters; decrease in size of wound, reduction of surrounding skin edema. Senior faculty will verify the assessment of wound healing.

Independent Variable Demographic variable: Age, Gender, Monthly household income Medical History: Blood profile, Pain Intervention: 1.Conventional dressings 2. Heparin Spray

Dependent Variable: Healing Time

2.9 Statistical Analyses: Statistical Package for Social Sciences (SPSS version 21) will be used for all statistical analyses.

Descriptive Statistics:

Descriptive statistics will be reported using mean and standard deviation for all continuous variables and frequencies and percentages for all categorical variables.

Inferential Statistics:

Mean wound healing time (recorded in days) between two intervention groups will be compared using Repeated measures ANOVA. p-value <0.05 will be considered as level of significance.

ELIGIBILITY:
Inclusion Criteria:

* • age between 18 to 55 years

  * both genders
  * non hypertensive patients
  * Hemoglobin levels more than 10 g/dl
  * Platelet count above 150 to 400 × 109/L
  * Wounds for more than 6 weeks
  * Any size of wound greater then 10*10 cm

Exclusion Criteria:

* • Hypertensive patients,

  * Bleeding tendencies (Disorder),
  * Immune-compromised,
  * Familial history of bleeding

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: general public
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-02 (Estimated)

PRIMARY OUTCOMES:
decrease in size of wound and decrease in surrounding skin edema | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: dr.faisal akhlaque, Study Director — dow university
Locations (1):
- Dr. Faraz, Karachi, Sindh, Pakistan

REFERENCES:
- [Derived] Adil F, Memon MA, Khan FAA, Awan A, Siddiqui SU, Piprani FZ, Zareen K. Efficacy of topical heparin spray on donor site wound healing after split thickness skin grafting. Sci Rep. 2025 Jul 30;15(1):27814. doi: 10.1038/s41598-025-95437-5. PMID 40738969